CLINICAL TRIAL: NCT00379938
Title: A Phase I/II Study of the Safety and Immunogenicity of a Recombinant Human Parvovirus B-19 Vaccine
Brief Title: B-19 Parvovirus Vaccine Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0078
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2009-02

CONDITIONS: Parvovirus B19 Infection
Keywords: Parvovirus B-19, Parvoviridae, vaccine
MeSH Terms: conditions — Erythema Infectiosum; Parvoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): 25 micrograms + MF59 (n=26)
  Interventions: Biological: VAI-VP705 (parvovirus B-19 vaccine); Biological: MF-59
- 3 (Experimental): 2.5 micrograms + MF59 (n=26)
  Interventions: Biological: VAI-VP705 (parvovirus B-19 vaccine); Biological: MF-59
- 4 (Placebo Comparator): saline (n=11)
  Interventions: Drug: Placebo
- 2 (Experimental): 25 micrograms alone (n=26)
  Interventions: Biological: VAI-VP705 (parvovirus B-19 vaccine)

INTERVENTIONS:
Biological: VAI-VP705 (parvovirus B-19 vaccine) — Recombinant human parvovirus B-19 capsids at dose levels: 25 micrograms of VAI-VP705 with and without MF59 adjuvant and 2.5 micrograms with MF59 adjuvant.
  Arms: 1; 2; 3
Drug: Placebo — Saline control
  Arms: 4
Biological: MF-59 — Adjuvant
  Arms: 1; 3

SUMMARY:
This study investigates the safety and effectiveness of a preventative vaccine for parvovirus B-19 infection. Eighty-nine healthy adults ages 18-49, whose blood tests negative for B-19, will be enrolled. Participants will be randomly chosen to receive 1 of 4 possible vaccine types: low dose of the vaccine and an adjuvant (substance which assists with transfer of medication to body); high dose of the vaccine alone; high dose of the vaccine and an adjuvant; or saline (substance containing no medication). Participants will receive 3 vaccinations over a 6 month period and will be followed for 6 additional months. Blood samples will be taken at months 1, 2, 6, 7 and 12 to determine if antibody, protein produced by the body's immune system that recognizes and helps fight infections, has been formed to the vaccine. These tests measure vaccine efficacy, i.e., determine if the vaccine induces immunity. All participants will be followed closely for safety throughout the study.

DETAILED DESCRIPTION:
This study is a Phase I/II randomized, placebo-controlled, double-blind clinical trial of the immunogenicity and safety of 2 dose levels of a recombinant human parvovirus B-19 vaccine (VAI-VP705). The vaccine is composed of viral capsids that incorporate 2 B-19 proteins (VP-1 and VP-2). There will be 3 sites participating in this study: Cincinnati Children's Hospital Medical Center, Baylor College of Medicine, and the University of Maryland School of Medicine. Eighty-nine parvovirus B-19 seronegative healthy adults 18-45 years old will be randomized to 1 of 4 groups: 2.5 mcg VAI-VP705 with the adjuvant MF59, 25 mcg with the adjuvant MF59, 25 mcg without the adjuvant MF59, or placebo (saline control). Each participant will receive 3 separate vaccinations (Months 0, 1, and 6) and will continue in the study for up to approximately 14 months. Study participants will be followed to evaluate safety and immune response. The primary study objective is to evaluate the safety of VAI-VP705 administered with and without MF59 adjuvant in healthy parvovirus B-19 seronegative adults. The secondary study objectives are to: evaluate the immunogenicity of primary and booster immunizations of 25 mcg of VAI VP705 with and without MF59 and 2.5 mcg with MF59; compare the antibody response of vaccine administered with MF59 at each of 2 doses, 2.5 and 25 mcg versus 25 mcg of vaccine administered without MF59; and evaluate the duration of the immune response 12 months after primary immunization. The primary endpoint is the number and percentage of study participants who experience any vaccine-associated adverse events or serious adverse events. The secondary endpoints include: the percentage of study participants who develop neutralizing antibody responses against parvovirus B-19 28 days following the last dose of vaccine; the percentage of study participants who maintain a neutralizing antibody titer at 12 months after primary immunization; the geometric mean antibody titers (as measured by enzyme-linked immunosorbent assay) by treatment group at 28 days and at 12 months after primary immunization; and the geometric mean neutralizing titers per treatment group at 28 days and at 12 months after primary immunization.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide informed consent;
* Must be between the ages of 18 to 45 at time of randomization;
* Must be in good health, as determined by vital signs (heart rate, blood pressure, respiration, and oral temperature), medical history, and a targeted physical examination based on medical history;
* Must have a negative serum pregnancy test at screening and negative urine pregnancy test prior to each vaccination (females);
* Must be medically or surgically sterile or agree to practice effective contraception (egg, oral contraceptives, diaphragm in combination with contraceptive jelly, cream, or foam; intrauterine contraceptive device; Depo-Provera; skin patch; vaginal ring or cervical cap) through 30 days after the final dose of study drug. Oral and hormonal contraceptives must be initiated at least 30 days prior to first dose of study drug and must continue through 30 days after the final dose of study drug;
* Must have a negative hepatitis B surface antigen (HBsAg) and hepatitis C virus (HCV) and HIV antibodies [by Enzyme-Linked Immunosorbent Assay (ELISA) and confirmed if positive by Western blot analysis [WBA]) prior to randomization);
* Must be seronegative for parvovirus B-19 by enzyme-linked immunosorbent assay [ELISA] prior to randomization.

Exclusion Criteria:

* Acute febrile illness (greater than or equal to 37.8 degrees Celcius/100 degrees Fahrenheit) within the 72 hours preceding the vaccination (vaccine may be deferred until resolved);
* Known exposure to persons with parvovirus B-19 (egg, fifth disease) within 6 weeks prior to randomization;
* Illness associated with parvovirus B-19 infection within 6 weeks prior to randomization;
* History of severe adverse reaction or allergy to any vaccine;
* Known or suspected allergies to vaccine constituents (egg, MF59);
* History of treatment with immunosuppressive drugs in the 30 days prior to enrollment (inhaled or topical corticosteroids are permitted) or for 28 days following last dose of vaccine;
* Treatment with blood or blood products within 3 months prior to enrollment or throughout the duration of the study;
* History of polyarthritis;
* A history or clinical manifestation of significant immunodeficiency, metabolic, pulmonary, cardiovascular, hepatic, renal, hematologic (including hereditary and hemolytic anemias), or gastrointestinal disorders;
* Clinically significant abnormal laboratory values at Screening including the following:

  1. Hgb <11.5 g/dL (females) or 12.5 g/dL (males); white blood cell (WBC) <4000/microliters; platelet count <135000/microliters;
  2. Alanine aminotransferase (ALT) or creatinine above the upper limits of normal.
* Any acute or chronic condition (including alcohol or drug abuse) that in the principal investigator's (PIs) opinion would limit the volunteer's ability to complete the study;
* Pregnant or breastfeeding;
* Receipt or planned receipt of any investigational drug, vaccine (exclusive of the vaccine under study), device or intervention within 30 days prior to randomization or through the 6 months following the last dose of study vaccine;
* Receipt of any licensed killed vaccine within 2 weeks before or after any dose of study vaccine;
* Receipt of any licensed, live, attenuated vaccine within 4 weeks before or after any dose of study vaccine;
* Any other condition that, in the opinion of the investigators, would place the subject at an unacceptable risk for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Number and percentage of study participants who experience any vaccine-associated AEs or SAEs. | Duration of study

SECONDARY OUTCOMES:
Geometric mean antibody titers (measured by Enzyme-Linked Immunosorbent Assay) by treatment group. | 28 days and 12 months after the primary immunization
Percentage of study participants who develop neutralizing antibody responses against parvovirus B-19. | 28 days following the last dose of vaccine
Percentage of study participants who maintain a neutralizing antibody titer. | 12 months after the primary immunization
Geometric mean neutralizing titer per treatment group. | 28 days and 12 months after the primary immunization

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas